CLINICAL TRIAL: NCT01611740
Title: Contribution of Computerized Real Time Analyses of Cardio-respiratory Signals to the Diagnosis of Infection in Preterm Infants
Brief Title: Contribution of Real Time Analyses of CARdio-RESpiratory Signals to the Diagnosis of Infection in PREterM Infants
Acronym: CARESS_PREMI
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00324-37
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Bacterial Infection
Keywords: Preterm infant; Bacterial infection; Diagnosis of proven or suspected bacterial infection
MeSH Terms: conditions — Bacterial Infections; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants: Telemonitoring system prototype developed by INSERM U-642
  Interventions: Procedure: Analysis of the heart rate and respiratory characteristics / Telemonitoring system prototype developed by INSERM U-642

INTERVENTIONS:
Procedure: Analysis of the heart rate and respiratory characteristics / Telemonitoring system prototype developed by INSERM U-642 — Telemonitoring system prototype developed by INSERM U-642 with analysis of :
  * the variability of the cardiac cycle duration ;
  * the variability of respiratory cycle amplitude and duration ;
  * and their relationships.

SUMMARY:
Hospital-acquired infections are common complications in preterm infants. The diagnosis has to be fast and accurate. Indeed, the early identification of a suspected infection is very important, since the early administration of antibiotics lowers the risk of septic shock and improves long term outcome in the infected newborns who survive. Besides, a high specificity in the diagnosis of infection allows for the reduction of inappropriate treatment and thus prevents the emergence of antibiotic resistance.

The aim of this study is to develop a computer-assisted diagnosis tool, based on the real time analysis of cardio-respiratory signals, to aid the neonatologist in the diagnosis of infection of the preterm infant, at the bedside.

DETAILED DESCRIPTION:
Hospital-acquired infections increase morbidity and mortality in the preterm infants. Early diagnosis of infection is difficult mainly due to the poor performance of clinical signs and to the need for invasive procedure to get blood tests. However, early administration of antibiotics lowers the risk of septic shock and improves long term outcome in the infected newborns who survive. Many clinical features have been described, associated with an ongoing infection but they are inconsistent, variable and nonspecific. Similarly, many invasive laboratory tests have been proposed for the diagnosis of infection in the newborn but they all need blood sampling and none has a good predictive value.

The combined analysis of the heart rate and respiratory characteristics appears to be a promising tool for the diagnosis of infection in the preterm infants. These signals are non-invasively recorded and their computerized real time analyses would allow for a continuous assessment of the risk of infection.

The main objective is to test the hypothesis that the analyses of the variability of the cardiac cycle duration, the variability of the respiratory cycle amplitude and duration, and their relationships, can significantly improve the performance of the diagnosis of late onset infection in the preterm infant at the bedside in neonatal units.

ELIGIBILITY:
Inclusion Criteria:

* preterm birth before < 32wks and > 24wks
* birth weight > 500g
* postnatal age> 3 days
* postconceptional age < 34wks
* parents information and collection of non-opposition

Exclusion Criteria:

* malformative syndrome
* severe neurological injury (IVH grade 4, cavitary periventricular leukomalacia, perinatal asphyxia post ischemia)

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm birth before < 32wks and > 24wks
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2012-05; Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Diagnosis of proven or suspected bacterial infection | Within the hospitalisation with an anticipated mean duration of 10 weeks
  The primary outcome will be the efficiency (area under curve, sensitivity, specificity, false-positive and false-negative) of the combined analysis of heart rate and respiratory characteristics for the diagnosis of proven or suspected bacterial infection.

SECONDARY OUTCOMES:
Inflammation without proven or suspected bacterial infection defined as follows: a 6 hours period with CRP> 5 mg/L not classified as proven or suspected bacterial infection. | Within the hospitalisation with an anticipated mean duration of 2 to 10 weeks
  We will investigate if this approach can discriminate an inflammation without proven or suspected bacterial infection defined as follows: a 6 hours period with CRP> 5 mg/L not classified as proven or suspected bacterial infection.
Periods of discomfort defined as at least two EDIN scores above 3 in a 6 hours period | Within the hospitalisation with an anticipated mean duration of 2 to 10 weeks
  The performance of a biomarker based on the computerized analyses of the cardiac and respiratory signals will also be tested for the detection of periods of discomfort defined as at least two EDIN scores above 3 in a 6 hours period.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD, PhD, Study Chair — Rennes University Hospital
Locations (3):
- France (3):
  - CHU Angers, Angers, Maine Et Loire
  - CHU de Lille, Lille
  - CHU de Rennes, Rennes